CLINICAL TRIAL: NCT05495321
Title: Therapeutic Effect of Interleukin-2 on Active Dermatomyositis: A Multicenter, Randomised, Double-blind, Placebo-controlled Trial
Brief Title: Interleukin-2 on Active Dermatomyositis
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Zhanguo Li, professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIMIL2
Record Dates: First submitted 2021-11-17; First posted 2022-08-10 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-dose IL-2 (Experimental): The first stage (double-blind treatment period): One million IU of IL-2 was injected subcutaneously once every other day for 12 weeks.
  The second stage (open treatment period): One million IU of IL-2 was injected subcutaneously once every other day for 12 weeks.
  Interventions: Drug: Interleukin-2
- Placebo (Placebo Comparator): The first stage (double-blind treatment period): Placebo was injected subcutaneously once every other day for 12 weeks.
  The second stage (open treatment period): One million IU of IL-2 was injected subcutaneously once every other day for 12 weeks.
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — low dose interleukin-2 injected subcutaneously, at a dose of 1 x 10~6 IU once every other day, for 6 months.
  Other Names: Recombinant Human Interleukin-2

SUMMARY:
The purpose of this paper is to explore the effect of low-dose IL-2 on refractory dermatomyositis and immunological indexes.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled, multicenter clinical trial was designed. Patients were treated with low-dose IL-2 regularly to explore its efficacy and safety. The improvement of clinical and laboratory indexes was evaluated. Changes of immune cell subsets and cytokines were monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (including 18 and 75 years old);
2. The diagnosis of dermatomyositis conforms to Bohan/Peter Recommendation in 1975 or EULAR/ACR Classification Standard in 2017.

   Active myositis was defined by baseline Manual Muscle Testing (MMT-8) no greater than 125/150 and at least two additional abnormal CSMs. To allow the enrolment of patients with active DM with a moderate to severe rash who may not meet the MMT-8 criterion noted above, patients with DM could be enrolled if their cutaneous VAS score on the Myositis Disease Activity Assessment Tool (MDAAT) was ≥3cm on the 10cm VAS scale and at least three of the five CSMs were abnormal (excluding the MMT-8).

   Abnormal CSMs include:
   * 1. patients global assessment (PGA), the minimum value of 10 cm visual analog scale (VAS) is 2.0 cm
   * 2. Physicians global assessment (PhGA), the minimum value on the 10 cm VAS scale is 2.0 cm
   * 3. Health Assessment Questionnaire (HAQ), with a minimum value of 0.25
   * 4. At least one muscle enzyme [including creatine kinase (CK), aldolase, lactate dehydrogenase (LDH), alanine aminotransferase (ALT) and aspartate aminotransferase (AST)] High, the lowest level is 1.3 x upper limit normal
   * 5. Global Extra-muscle Disease Activity Score, with a minimum of 1.0 cm on the 10 cm VAS scale [This measure is a comprehensive assessment by the physician based on an assessment of the physique, skin, bone, gastrointestinal, lung and heart scale activity scores,named Myositis Disease Activity Assessment Tool (MDAAT)].
   * 6. Manual Muscle Testing (MMT-8) no greater than 125/150.
3. The dose of glucocorticoid (equivalent to prednisone) was less than 0.5mg/kg/d within 4 weeks before joining the group, and/or there were no new immunosuppressants (cyclophosphamide, mycophenolate mofetil, cyclosporine, tacrolimus, azathioprine, methotrexate, etc.) within 12 weeks, and the dose was stable for 4 weeks.
4. Voluntary signing of informed consent: When participating in the trial, the patient must be given a written notice of consent, and hope that the patient can comply with the requirements of the study follow-up plan and other protocols.
5. Agree to adopt effective contraceptive measures during the study period (women of childbearing age).

Exclusion Criteria:

Any subject meeting any of the following criteria should be excluded:

1. Received intravenous glucocorticoid (> 1 mg/kg/d) within 4 weeks;
2. Serious complications: including (1). heart failure (≥ NYHA III); (2). renal insufficiency (creatinine clearance rate ≤30 ml/min); (3). liver insufficiency (excluding serum ALT or AST caused by dermatomyositis, or total bilirubin greater than normal upper limit), (4). hemoglobin < 80g/L, E. platelet count < 60.
3. Dermatomyositis patients with other connective tissue diseases or tumors;
4. Allergic constitution or allergic to multiple drugs;
5. Those who are in the period of acute and chronic infection (including but not limited to hepatitis, pneumonia, bacteremia, pyelonephritis, Epstein-Barr virus, tuberculosis infection), or are hospitalized for infection, or use intravenous antibiotics to treat infection 2 months before the first treatment, or have a history of active tuberculosis in the past;
6. Those who are positive for hepatitis B surface antigen or hepatitis C antibody;
7. Persons with mental illness or other reasons who cannot cooperate with treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving minimal improvement (TIS≥20). | week 12
  The primary outcome will be to compare the proportion of subjects achieving minimal improvement (TIS≥20). The TIS (total improvement score) is the sum of all 6 improvement scores associated with the change in each core set measure. A total improvement score of ≥20 represents minimal improvement, a score of ≥40 represents moderate improvement, and a score of ≥60 represents major improvement.

SECONDARY OUTCOMES:
MMT-8 (Manual Muscle Testing), (potential score 0 - 80); | week12 and 24
  MMT-8 is a set of 8 designated muscles tested unilaterally; test on right side (use left side if right side cannot be tested). Higher scores mean a better outcome.
CDASI activity score (cutaneous dermatomyositis disease area and severity index), (potential score 0-100 for cutaneous dermatomyositis disease area and 0-32 for severity index); | week12 and 24
  The CDASI is a clinician-scored single page instrument that separately measures activity and damage in the skin of DM patients for use in clinical practice or clinical/therapeutic studies. Higher scores mean a worse outcome.
Physician's Global Disease Activity VAS, (potential score 0 - 10); | week12 and 24
  Physician's Global Disease Activity (10 cm VAS assessing global disease activity from "No evidence of disease activity" to "Extremely active or severe disease activity"; Disease Activity being defined as potentially reversible pathology or physiology resulting from the myositis). Higher scores mean a worse outcome.
Patient's Global Disease Activity VAS, (potential score 0 - 80); | week 12 and 24
  Patient's Global Disease Activity (10 cm VAS assessing global disease activity from "No evidence of disease activity" to "Extremely active or severe disease activity"; Disease Activity being defined as potentially reversible pathology or physiology resulting from the myositis). Higher scores mean a worse outcome.
Health assessment question, (potential score 0 - 3); | week 12 and 24
  Patients reported how their illness affects their ability to function in daily life , Higher scores mean a better outcome.
Myositis disease activity assessment tool (MDAAT) - 2005, VERSION 2 | week 12 and 24
  This is a combined tool that captures the physician's assessment of disease activity of various organ systems using (1) the 0-4 scale described below and (2) a visual analog scale (VAS) [potential score 0 - 10]. Please assess the clinical features (items 1-26) of each organ system. Higher scores mean a worse outcome.
CD4 T cells | week 12 and 24
  number and proportion of CD4 T cells in peripheral blood.
Serum cytokines | week 12 and 24
  concentration of serum cytokines
glucocorticoid dosage | week 12 and 24
  Daily dosage of glucocorticoid
Rate of Participants with adverse effects associated with experimental drugs | up to 24 weeks
  Adverse effects include fever, rash, abnormal liver function, rate of new-onset infection and any abnormal measures associated with low-dose IL-2 therapy.
Proportion of subjects meeting the definition of improvement (DOI) | week12 and 24
  The DOI for this trial is a composite utilizing the six CSM: 3 of 6 CSM improved by ≥ 20%, with no more than 2 CSM worsening by ≥25% (a worsening measure cannot be the MMT).
Number of subjects achieving minimal improvement (TIS≥20). | week 24
  The primary outcome will be to compare the proportion of subjects achieving minimal improvement (TIS≥20). The TIS (total improvement score) is the sum of all 6 improvement scores associated with the change in each core set measure. A total improvement score of ≥20 represents minimal improvement, a score of ≥40 represents moderate improvement, and a score of ≥60 represents major improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Zhanguo Li, Study Director — Peking University People's Hospital
Locations (1):
- Peking university people's hospital, Beijing, Beijing Municipality, China